CLINICAL TRIAL: NCT06968091
Title: Effect of Trendelenburg Positioning on Anesthesia-Induced Hypotension in Elderly Patients: A Randomized Controlled Clinical Trial
Brief Title: Effect of Trendelenburg Positioning on Anesthesia-Induced Hypotension in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Gu Bin, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-2025-478
Record Dates: First submitted 2025-05-03; First posted 2025-05-13 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Hypotension on Induction; Old Age
MeSH Terms: interventions — Head-Down Tilt

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The anesthesiologists do not implement the blinding method for the patient grouping, while the physicians conducting the postoperative follow-up implement the blinding method for the grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Trendelenburg Position Group (Experimental)
  Interventions: Other: Trendelenburg position
- The Supine Horizontal Position Group (Placebo Comparator)
  Interventions: Other: Supine Horizontal Position

INTERVENTIONS:
Other: Trendelenburg position — After the loss of consciousness during general anesthesia, the 10° Trendelenburg position is adopted.
  Arms: The Trendelenburg Position Group
Other: Supine Horizontal Position — After the loss of consciousness during general anesthesia, the Supine Horizontal Position is adopted.
  Arms: The Supine Horizontal Position Group

SUMMARY:
This study investigated the effect of Trendelenburg position on preventing post-induction hypotension in elderly patients undergoing abdominal surgery with general anesthesia. The patients will receive the 10° Trendelenburg position or supine position during anesthesia induction. The primary outcome is the area under a mean arterial pressure (MAP) below 65 mm Hg within the first 15 minutes during anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65-90 years
* scheduled for abdominal surgery with general anesthesia
* expected to have continuous radial arterial pressure monitoring
* American Society of Anesthesiologists (ASA) physical status I to III

Exclusion Criteria:

* contraindications or failure of radial arterial catheterization
* expected possible difficult airway
* non-sinus rhythm
* increased intracranial pressure
* patients at high risk of regurgitation or aspiration
* inability to provide consent

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The area under the curve of the mean arterial pressure being lower than 65 mmHg | within 15 minutes after anesthesia induction

SECONDARY OUTCOMES:
The area under the curve of the mean arterial pressure being lower than 60 mmHg | within 15 minutes after anesthesia induction
The area under the curve of the mean arterial pressure being lower than 50 mmHg | within 15 minutes after anesthesia induction
The area under the curve of the mean arterial pressure being lower than 40 mmHg | within 15 minutes after anesthesia induction
The duration during which the Mean Arterial Pressure (MAP) is less than 65 mmHg | within 15 minutes after anesthesia induction
The duration during which the Mean Arterial Pressure (MAP) is less than 60 mmHg | within 15 minutes after anesthesia induction
The duration during which the Mean Arterial Pressure (MAP) is less than 50 mmHg | within 15 minutes after anesthesia induction
The duration during which the Mean Arterial Pressure (MAP) is less than 40 mmHg | within 15 minutes after anesthesia induction
The usage of vasoactive drugs | within 15 minutes after anesthesia induction and during the whole process of the surgery
  The vasoactive drugs are selected from the following according to the protocol: phenylephrine, ephedrine, norepinephrine, and epinephrine.
The lowest mean arterial pressure | within 15 minutes after anesthesia induction
the postoperative complications | within 30 days after surgery
  The complications are assessed using the Claviene-Dindo score.
the postoperative recovery | on postoperative day 1
  The postoperative recovery is assessed using the quality of recovery-15 questionnaire (QoR-15) .The QoR-15 has 15 questions. Each question is rated on a 10-point scale, ranging from 0 (none of the time or poor) to 10 (all of the time or excellent). The maximum score (best recovery) is 150.
Length of hospital stay after surgery | through study completion, an average of 3-15 days
The time duration required to complete endotracheal intubation | through study completion, an average of 10-60 s
The incidence of refractory hypotension | within 15 minutes after anesthesia induction
  If either of the following two definitions is met, it is considered refractory hypotension:
  1. During the anesthesia induction period, the total administered dosage exceeds the maximum dose, and the patient's hypotension does not recover. The maximum usage dose of ephedrine is 0.5 mg/kg (ideal body weight), and the maximum usage dose of phenylephrine is 8 μg/kg (ideal body weight).
  2. When two or more vasoactive drugs are used, the systolic blood pressure is less than 80 mmHg or the mean blood pressure is less than 65 mmHg continuously for more than 5 minutes.
The number of attempts at tracheal intubation | through study completion, an average of 1-2times
The dosage of propofol during the anesthesia induction period | within 15 minutes after anesthesia induction
The dosage of remifentanil during the anesthesia induction period | within 15 minutes after anesthesia induction
The VIDIAC score of the video laryngoscope. | through study completion, an average of -1~1 points
  The VIDIAC score is comprised of: E, the interaction between the blade tip and epiglottis; V, the best view of the vocal cords from the blade camera; and A, enlargement of the arytenoids. The score range of the VIDIAC score is from -1 to 5 points. The VIDIAC score classification is as follows: Easy, with a score of -1 or 0; Moderate, with a score of 1; Difficult, with a score of 2; Severe, with a score of ≥3.
The usage of other medications during the anesthesia induction period | within 15 minutes after anesthesia induction
  The usage of medications other than propofol, remifentanil, phenylephrine, ephedrine, norepinephrine, and epinephrine.
The area under the curve of the mean arterial pressure being lower than 65 mmHg | within 20 minutes after anesthesia induction
The pulse pressure variation rate after mechanical ventilation. | At the 1st, 3rd, 5th and 10th minutes after tracheal intubation
The peak airway pressure after mechanical ventilation. | At the 1st minutes after tracheal intubation
The infusion volume of crystalloid solution during the induction period. | within 15 minutes after anesthesia induction
Arterial systolic pressure after anesthesia induction | At the 1st, 2nd, 3rd, 4th, 5th, 6th, 7th, 8th, 9th, 10th, 11th, 12th, 13th, 14th, 15th, 16th, 17th, 18th, 19th and 20th minutes after anesthesia induction.
  The monitor records continuous arterial blood pressure data at intervals of 1 second.
Arterial diastolic pressure after anesthesia induction | At the 1st, 2nd, 3rd, 4th, 5th, 6th, 7th, 8th, 9th, 10th, 11th, 12th, 13th, 14th, 15th, 16th, 17th, 18th, 19th and 20th minutes after anesthesia induction.
  The monitor records continuous arterial blood pressure data at intervals of 1 second.
Mean arterial pressure after anesthesia induction | At the 1st, 2nd, 3rd, 4th, 5th, 6th, 7th, 8th, 9th, 10th, 11th, 12th, 13th, 14th, 15th, 16th, 17th, 18th, 19th and 20th minutes after anesthesia induction.
  The monitor records continuous arterial blood pressure data at intervals of 1 second.
Heart rate after anesthesia induction | At the 1st, 2nd, 3rd, 4th, 5th, 6th, 7th, 8th, 9th, 10th, 11th, 12th, 13th, 14th, 15th, 16th, 17th, 18th, 19th and 20th minutes after anesthesia induction.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang cancer hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
We will share data on ClinicalTrials.gov, and data sharing will be always available.
Supporting Information: Study Protocol, Analytic Code
Time Frame: starting about 6 months after publication